CLINICAL TRIAL: NCT03194087
Title: the Study on Difference Prognostic for Low Parathyroid Hormone Levels and Severe Secondary Hyperparathyroidism in Hemodialysis Patients
Brief Title: the Study on Prognostic for Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wenhu Liu, Professor, Beijing Friendship Hospital
Other Study IDs: 2016-P2-044-01
Record Dates: First submitted 2017-05-31; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Secondary Hyperparathyroidism; Low parathyroid hormone; Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Results from KDOQI guidelines, parathyroid hormone (PTH) level within target range is 150-300pg/ml. Both lower PTH levels and higher PTH levels were associated with higher risk of all-cause mortality. However, in out of target range, it is still unknown which mortality higher. so, in this prospective, observational clinical trial study. the investigators will observe the mortality and cardiovascular incidence rate between SHPT(>800pg/ml) and low serum PTH levels(<60pg/ml). Both two groups of patients will receive a reasonable treatment according to the suggestions in K/DOQI guidelines.

DETAILED DESCRIPTION:
It is common that the abnormalities in parathyroid hormone (PTH) levels appear in patients with moderate and advanced chronic kidney diseases (CKD). CKD-mineral and bone disorder (CKD-MBD), manifested by the serum calcium (Ca), phosphorus (P), and parathyroid hormone (PTH) levels, and other abnormalities such as vitamin D metabolism and bone turnover etc, contribute to the increased morbidity and mortality in patients on maintenance dialysis.

Results from KDOQI guidelines, indicated that an increased mortality risk was associated with high parathyroid hormone (PTH) levels, if the PTH levels >600pg/ml, it means severe secondary hyperparathyroidism, it have been shown to contribute to alterations of arterial structure and function and associated with cardiovascular (CV), calcifications, CV events, and death.

In most patients, SHPT can be successfully controlled by dialysis and supplements of calcium and vitamin D. but Results from several studies, the severe secondary hyperparathyroidism can't be control by medical treatment or hemodialysis, about 15% of patients after 10 years and 38% of patients after 20 years of dialysis need parathyroidectomy. total parathyroidectomy(tPTX) is the best Surgical approach. tPTX seems to be associated to a lower relapse rate but higher percentage of hypoparathyroidism. But it may cause the patient in low parathyroid hormone status.

It is well known that at present, a high proportion of patients receiving dialysis therapy have relatively low serum PTH levels. In parallel, the observation that CV calcifications are more prevalent in patients undergoing dialysis who have low serum PTH levels than in those with normal or moderately elevated levels, in association with low-turnover bone disease, this condition favors mineral deposition in vascular and other soft tissues instead of bone. Results from several studies, all of them reported an increase in CV mortality risk in patients with low PTH levels.

Nonetheless, consistent evidence associating Compare SHPT with low serum PTH levels which mortality rate is higher in patients undergoing dialysis is still lacking. so, in this prospective, observational clinical trial study. the investigators will observe the mortality and CV incidence rate between SHPT and low serum PTH levels. the investigators detect the iPTH levels of all the patients in the investigators' blood purification center. The patients whose iPTH are Less than 300pg/ml and more than the 800pg/ml are chosen to involve in this study. According to PTH levels The patients will be divided into two groups. Both two groups of patients will receive a reasonable treatment according to the suggestions in K/DOQI guidelines. Then, all of the patients will be followed for 24 months to compare the rate of cardiovascular and cerebrovascular events and mortality in each group.

ELIGIBILITY:
Inclusion Criteria:

1. patients with age between 18-75 years.
2. patients in hemodialysis, whose iPTH is below 300pg/ml or above 800pg/ml.

Exclusion Criteria:

1. primary or tertiary hyperparathyroidism(hyperparathyroidism after kidney transplantation).
2. pregnant or lactating woman.
3. patients with severe liver disease and abnormal blood clotting mechanism.
4. patients with chronic wasting disease.
5. patients whose concurrent illnesses,disability,or geographical residence would hamper attendance at required study visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. patients with age between 18-75 years.
  2. patients in hemodialysis, whose iPTH is below 300pg/ml or above 800pg/ml.
Sampling Method: Probability Sample
Enrollment: 827 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 24 months
  all of the patients will be followed for 24 months to compare the all-cause mortality.

SECONDARY OUTCOMES:
the rate of cardiovascular and cerebrovascular events. | 24 months
  all of the patients will be followed for 24 months to compare the rate of cardiovascular and cerebrovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: WenHu Liu, doctor, Study Chair — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No